CLINICAL TRIAL: NCT04863768
Title: Molecular Profiling of Colorectal Cancer: A Translational Research Study With a Next Generation Sequencing Panel.
Brief Title: Molecular Profiling of Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: TR6N/19
Record Dates: First submitted 2021-03-12; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-03

CONDITIONS: Colorectal Cancer; Colon Cancer; Colon Adenocarcinoma
Keywords: Colon; Translational research; Gene panel
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Formalin-Fixed-Paraffin-Embedded (FFPE) tumor tissue blocks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Gene panel — comprehensive cancer gene panel targeting regions in 37 clinically relevant cancer genes in FFPE tumor tissue blocks

SUMMARY:
In this translational research study, Formalin-Fixed-Paraffin-Embedded (FFPE) tumor tissue blocks from patients with early-stage (II-III) colorectal cancer will be assessed for a comprehensive cancer gene panel from NIPD Genetics (https://www.nipd.com/) targeting regions in 37 clinically relevant cancer genes.

The colorectal cancer panel includes an extended list of clinically relevant genes, designed to target clinically actionable and clinically significant mutations that will provide physicians with genetic information regarding a) prediction of the patient's response to targeted therapy, b) prognosis, that is, prediction of clinical outcome, c) diagnosis and molecular classification of colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Surgically resected early-stage (II-III) colorectal cancer
* Availability of biological material

Exclusion Criteria:

* Metastatic disease (stage IV) at initial diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent surgical resection of early-stage (II-III) colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2006-01-01 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
association between gene mutational status and overall survival | 24 months
  the time from diagnosis to the date of death (from any cause). Alive patients and patients lost to follow-up will be censored at the date of last follow-up
association between gene mutational status and disease-free survival | 24 months
  the time from colorectal cancer diagnosis to the first date of documented disease progression, death or last contact, whichever occurs first

SECONDARY OUTCOMES:
Descriptives | 24 months
  Association of any gene mutation tumor pathological stages.
Descriptives | 24 months
  Association of any gene mutation tumor budding.
Descriptives | 24 months
  Association of any gene mutation with microstatellite instability.

CONTACTS AND LOCATIONS:
Overall Officials: George Fountzilas, Prof, Study Chair — Hellenic Cooperative Oncology Group
Locations (1):
- Hellenic Cooperative Oncology Group, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dekker E, Tanis PJ, Vleugels JLA, Kasi PM, Wallace MB. Colorectal cancer. Lancet. 2019 Oct 19;394(10207):1467-1480. doi: 10.1016/S0140-6736(19)32319-0. PMID 31631858
- [Background] Seufferlein T, Simoes C, Kude F, Ettrich TJ. Molecular Approaches to Metastatic Colorectal Cancer: Better Diagnosis - Better Treatment? Visc Med. 2019 Aug;35(4):259-264. doi: 10.1159/000500617. Epub 2019 Jul 11. PMID 31602389
- [Background] Khan K, Valeri N, Dearman C, Rao S, Watkins D, Starling N, Chau I, Cunningham D. Targeting EGFR pathway in metastatic colorectal cancer- tumour heterogeniety and convergent evolution. Crit Rev Oncol Hematol. 2019 Nov;143:153-163. doi: 10.1016/j.critrevonc.2019.09.001. Epub 2019 Sep 7. PMID 31678702
- [Background] Cohen R, Rousseau B, Vidal J, Colle R, Diaz LA Jr, Andre T. Immune Checkpoint Inhibition in Colorectal Cancer: Microsatellite Instability and Beyond. Target Oncol. 2020 Feb;15(1):11-24. doi: 10.1007/s11523-019-00690-0. PMID 31786718
- [Background] Caputo F, Santini C, Bardasi C, Cerma K, Casadei-Gardini A, Spallanzani A, Andrikou K, Cascinu S, Gelsomino F. BRAF-Mutated Colorectal Cancer: Clinical and Molecular Insights. Int J Mol Sci. 2019 Oct 28;20(21):5369. doi: 10.3390/ijms20215369. PMID 31661924
- [Background] Oh HH, Joo YE. Novel biomarkers for the diagnosis and prognosis of colorectal cancer. Intest Res. 2020 Apr;18(2):168-183. doi: 10.5217/ir.2019.00080. Epub 2019 Nov 30. PMID 31766836
- [Background] De Roock W, Claes B, Bernasconi D, De Schutter J, Biesmans B, Fountzilas G, Kalogeras KT, Kotoula V, Papamichael D, Laurent-Puig P, Penault-Llorca F, Rougier P, Vincenzi B, Santini D, Tonini G, Cappuzzo F, Frattini M, Molinari F, Saletti P, De Dosso S, Martini M, Bardelli A, Siena S, Sartore-Bianchi A, Tabernero J, Macarulla T, Di Fiore F, Gangloff AO, Ciardiello F, Pfeiffer P, Qvortrup C, Hansen TP, Van Cutsem E, Piessevaux H, Lambrechts D, Delorenzi M, Tejpar S. Effects of KRAS, BRAF, NRAS, and PIK3CA mutations on the efficacy of cetuximab plus chemotherapy in chemotherapy-refractory metastatic colorectal cancer: a retrospective consortium analysis. Lancet Oncol. 2010 Aug;11(8):753-62. doi: 10.1016/S1470-2045(10)70130-3. Epub 2010 Jul 8. PMID 20619739
- [Background] Strimpakos A, Pentheroudakis G, Kotoula V, De Roock W, Kouvatseas G, Papakostas P, Makatsoris T, Papamichael D, Andreadou A, Sgouros J, Zizi-Sermpetzoglou A, Kominea A, Televantou D, Razis E, Galani E, Pectasides D, Tejpar S, Syrigos K, Fountzilas G. The prognostic role of ephrin A2 and endothelial growth factor receptor pathway mediators in patients with advanced colorectal cancer treated with cetuximab. Clin Colorectal Cancer. 2013 Dec;12(4):267-274.e2. doi: 10.1016/j.clcc.2013.07.001. Epub 2013 Sep 17. PMID 24050852
- [Background] Pentheroudakis G, Kotoula V, De Roock W, Kouvatseas G, Papakostas P, Makatsoris T, Papamichael D, Xanthakis I, Sgouros J, Televantou D, Kafiri G, Tsamandas AC, Razis E, Galani E, Bafaloukos D, Efstratiou I, Bompolaki I, Pectasides D, Pavlidis N, Tejpar S, Fountzilas G. Biomarkers of benefit from cetuximab-based therapy in metastatic colorectal cancer: interaction of EGFR ligand expression with RAS/RAF, PIK3CA genotypes. BMC Cancer. 2013 Feb 2;13:49. doi: 10.1186/1471-2407-13-49. PMID 23374602
- [Background] Pagani F, Randon G, Guarini V, Raimondi A, Prisciandaro M, Lobefaro R, Di Bartolomeo M, Sozzi G, de Braud F, Gasparini P, Pietrantonio F. The Landscape of Actionable Gene Fusions in Colorectal Cancer. Int J Mol Sci. 2019 Oct 25;20(21):5319. doi: 10.3390/ijms20215319. PMID 31731495
- [Background] Itatani Y, Kawada K, Yamamoto T, Sakai Y. Resistance to Anti-Angiogenic Therapy in Cancer-Alterations to Anti-VEGF Pathway. Int J Mol Sci. 2018 Apr 18;19(4):1232. doi: 10.3390/ijms19041232. PMID 29670046
- [Background] Pentheroudakis G, Mavroeidis L, Papadopoulou K, Koliou GA, Bamia C, Chatzopoulos K, Samantas E, Mauri D, Efstratiou I, Pectasides D, Makatsoris T, Bafaloukos D, Papakostas P, Papatsibas G, Bombolaki I, Chrisafi S, Kourea HP, Petraki K, Kafiri G, Fountzilas G, Kotoula V. Angiogenic and Antiangiogenic VEGFA Splice Variants in Colorectal Cancer: Prospective Retrospective Cohort Study in Patients Treated With Irinotecan-Based Chemotherapy and Bevacizumab. Clin Colorectal Cancer. 2019 Dec;18(4):e370-e384. doi: 10.1016/j.clcc.2019.07.007. Epub 2019 Jul 15. PMID 31402291
- [Background] Pentheroudakis G, Kotoula V, Fountzilas E, Kouvatseas G, Basdanis G, Xanthakis I, Makatsoris T, Charalambous E, Papamichael D, Samantas E, Papakostas P, Bafaloukos D, Razis E, Christodoulou C, Varthalitis I, Pavlidis N, Fountzilas G. A study of gene expression markers for predictive significance for bevacizumab benefit in patients with metastatic colon cancer: a translational research study of the Hellenic Cooperative Oncology Group (HeCOG). BMC Cancer. 2014 Feb 20;14:111. doi: 10.1186/1471-2407-14-111. PMID 24555920
- [Background] Koutras AK, Antonacopoulou AG, Eleftheraki AG, Dimitrakopoulos FI, Koumarianou A, Varthalitis I, Fostira F, Sgouros J, Briasoulis E, Bournakis E, Bafaloukos D, Bompolaki I, Galani E, Kalogeras KT, Pectasides D, Fountzilas G, Kalofonos HP. Vascular endothelial growth factor polymorphisms and clinical outcome in colorectal cancer patients treated with irinotecan-based chemotherapy and bevacizumab. Pharmacogenomics J. 2012 Dec;12(6):468-75. doi: 10.1038/tpj.2011.37. Epub 2011 Aug 16. PMID 21844885
- [Background] Stratton MR, Campbell PJ, Futreal PA. The cancer genome. Nature. 2009 Apr 9;458(7239):719-24. doi: 10.1038/nature07943. PMID 19360079
- [Background] Chin L, Gray JW. Translating insights from the cancer genome into clinical practice. Nature. 2008 Apr 3;452(7187):553-63. doi: 10.1038/nature06914. PMID 18385729
- [Background] Forbes SA, Beare D, Boutselakis H, Bamford S, Bindal N, Tate J, Cole CG, Ward S, Dawson E, Ponting L, Stefancsik R, Harsha B, Kok CY, Jia M, Jubb H, Sondka Z, Thompson S, De T, Campbell PJ. COSMIC: somatic cancer genetics at high-resolution. Nucleic Acids Res. 2017 Jan 4;45(D1):D777-D783. doi: 10.1093/nar/gkw1121. Epub 2016 Nov 28. PMID 27899578
- [Background] Cancer Genome Atlas Research Network; Weinstein JN, Collisson EA, Mills GB, Shaw KR, Ozenberger BA, Ellrott K, Shmulevich I, Sander C, Stuart JM. The Cancer Genome Atlas Pan-Cancer analysis project. Nat Genet. 2013 Oct;45(10):1113-20. doi: 10.1038/ng.2764. PMID 24071849
- [Background] Landrum MJ, Lee JM, Riley GR, Jang W, Rubinstein WS, Church DM, Maglott DR. ClinVar: public archive of relationships among sequence variation and human phenotype. Nucleic Acids Res. 2014 Jan;42(Database issue):D980-5. doi: 10.1093/nar/gkt1113. Epub 2013 Nov 14. PMID 24234437
- [Background] Jennings LJ, Arcila ME, Corless C, Kamel-Reid S, Lubin IM, Pfeifer J, Temple-Smolkin RL, Voelkerding KV, Nikiforova MN. Guidelines for Validation of Next-Generation Sequencing-Based Oncology Panels: A Joint Consensus Recommendation of the Association for Molecular Pathology and College of American Pathologists. J Mol Diagn. 2017 May;19(3):341-365. doi: 10.1016/j.jmoldx.2017.01.011. Epub 2017 Mar 21. PMID 28341590
- [Background] Koumbaris G, Kypri E, Tsangaras K, Achilleos A, Mina P, Neofytou M, Velissariou V, Christopoulou G, Kallikas I, Gonzalez-Linan A, Benusiene E, Latos-Bielenska A, Marek P, Santana A, Nagy N, Szell M, Laudanski P, Papageorgiou EA, Ioannides M, Patsalis PC. Cell-Free DNA Analysis of Targeted Genomic Regions in Maternal Plasma for Non-Invasive Prenatal Testing of Trisomy 21, Trisomy 18, Trisomy 13, and Fetal Sex. Clin Chem. 2016 Jun;62(6):848-55. doi: 10.1373/clinchem.2015.252502. Epub 2016 Apr 26. PMID 27117469